CLINICAL TRIAL: NCT07261241
Title: NANT 2021-02: A Randomized Phase 2 Study of 131I-MIBG With Vorinostat VS. 131I-MIBG With Dinutuximab vs. 131I-MIBG With Dinutuximab and Vorinostat for Relapsed or Refractory Neuroblastoma
Brief Title: NANT 2021-02: Randomized MIBG With Vorinostat/Dinutuximab/Vorinostat + Dinutuximab
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: New Approaches to Neuroblastoma Therapy Consortium (Other)
Collaborators: United Therapeutics (Industry); Jubilant DraxImage Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NANT 2021-02
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — 3-Iodobenzylguanidine; dinutuximab; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: 131I-MIBG + vorinostat (Experimental): Patients assigned to Arm A will receive vorinostat orally once daily on Days 0 to 13 at a dose of 180 mg/m2/dose (maximum dose 400 mg). Patients will receive 131I-MIBG 18 mCi/kg (maximum dose 1200 mCi) on Day 1 and autologous stem cell infusion on Day 15 (plus 2 days or minus 1 day, hereafter abbreviated as +2/-1 days). There must be at least 24 hours between the last dose of vorinostat and stem cell infusion.
  Disease evaluation is to occur between days 50-60. The time interval between performing end of Course 1 disease evaluation and administration of Course 2 131I-MIBG is not to exceed 4 weeks.
  Interventions: Drug: Radiation: 131I-MIBG; Drug: Vorinostat
- Arm B: 131I-MIBG + dinutuximab (Experimental): Patients assigned to Arm B will receive 18 mCi/kg (maximum dose 1200 mCi) 131I-MIBG on Day 1 and autologous stem cell infusion on Day 15 (+2/-1 days). Dinutuximab 17.5 mg/m2/day is given intravenously on Days 8-11 and 29-32 of therapy.
  Disease evaluation is to occur between Days 50-60. In case of treatment delays with dinutuximab during Course 1, the time interval between performing end of Course 1 disease evaluation and administration of Course 2 131I-MIBG is not to exceed 4 weeks.
  Interventions: Drug: Radiation: 131I-MIBG; Drug: Dinutuximab
- Arm C: 131I-MIBG + vorinostat + dinutuximab (Experimental): Patients assigned to Arm C will receive vorinostat 180 mg/m2/dose (maximum dose 400 mg) on Days 0 to 13, 131I-MIBG 18 mCi/kg (maximum dose 1200 mCi) on Day 1. Dinutuximab 17.5 mg/m2/day is given intravenously on Days 8-11 and 29-32 of therapy.
  Disease evaluation is to occur between Days 50-60. In case of treatment delays with dinutuximab during Course 1, the time interval between performing end of Course 1 disease evaluation and administration of Course 2 131I-MIBG is not to exceed 4 weeks.
  Interventions: Drug: Radiation: 131I-MIBG; Drug: Dinutuximab; Drug: Vorinostat

INTERVENTIONS:
Drug: Radiation: 131I-MIBG — Patients will receive 131I-MIBG 18 mCi/kg (maximum dose 1200 mCi) on Day 1
  Other Names: Iobenguane I 131
Drug: Dinutuximab — Dinutuximab 17.5 mg/m2/day is given intravenously on Days 8-11 and 29-32 of therapy
  Other Names: Chimeric Monoclonal Antibody 14.18; Chimeric MOAB 14.18; human/murine anti-GD2 monoclonal antibody; chimeric anti-GD2; chimeric mAb 14.18; ch14.18; Unituxin
  Arms: Arm B: 131I-MIBG + dinutuximab; Arm C: 131I-MIBG + vorinostat + dinutuximab
Drug: Vorinostat — Vorinostat will be given on days 0-13 at a dose of 180 mg/m2/dose (maximum dose 400 mg).
  Other Names: Zolinza
  Arms: Arm A: 131I-MIBG + vorinostat; Arm C: 131I-MIBG + vorinostat + dinutuximab

SUMMARY:
Patients will then be randomized at study entry to one of three treatment arms. Patients on Arm A will receive a single treatment course with 131I-MIBG with vorinostat. Patients on Arm B will receive a single treatment course with 131I-MIBG and dinutuximab. Patients on Arm C will receive a single treatment course with 131I-MIBG with dinutuximab + vorinostat. After this course of treatment, we will check to see your response and then check to see how you are doing over time. All patients may choose to proceed to a second course of the same treatment if they and their physician feel healthy enough to do so. Approximately 118 patients will be receiving therapy on this trial.

DETAILED DESCRIPTION:
The proposed study is a 3-arm randomized, pick-the-winner, phase 2 trial designed to identify the optimal combination 131I-MIBG treatment regimen for further study. The three treatment arms are 131I-MIBG + vorinostat; 131I-MIBG + dinutuximab; and 131I-MIBG + dinutuximab + vorinostat. Objective response rate following a single course of therapy will be the primary endpoint driving selection of the regimen to move forward into future studies.

ELIGIBILITY:
Inclusion Criteria:

Age Patients must be ≥ 1 year and < 30 years of age at the time of study registration.

Diagnosis Patients must have a diagnosis of neuroblastoma or ganglioneuroblastoma nodular subtype either by histologic verification of neuroblastoma and/or demonstration of tumor cells in the bone marrow with increased urinary catecholamines.

Disease Risk Group Patients must have high risk neuroblastoma according to COG risk classification at the time of study registration. Patients who were initially considered low or intermediate risk, but then reclassified as high risk are also eligible.

Response to Prior Therapy (using INRC definitions)

Patients must have at least ONE of the following:

* Recurrent/progressive disease after the diagnosis of high risk neuroblastoma at any time prior to enrollment - regardless of response to frontline therapy. (Note that this excludes patients initially considered low or intermediate risk that progressed to high risk disease but have not progressed after the diagnosis of high risk neuroblastoma).
* If no prior history of recurrent/progressive disease since the diagnosis of high risk neuroblastoma,
* Refractory disease: A best overall response of no response/stable disease since diagnosis of high risk neuroblastoma AND after at least 4 courses of induction therapy.
* Persistent disease: A best overall response of minor response since diagnosis of high risk neuroblastoma AND after at least 4 courses of induction therapy:

  i. If a patient with persistent disease has 3 or more MIBG avid sites (including all soft tissue and/or bone lesions) OR a Curie Score of ≥ 3, then no biopsy is required for eligibility.

ii. If a patient with persistent disease has only 1 or 2 MIBG avid sites (including all soft tissue and/or bone lesions) then biopsy confirmation of neuroblastoma and/or ganglioneuroblastoma in at least one MIBG avid site (bone marrow, bone, or soft tissue) present at the time of registration is required. Bone and/or soft tissue lesions may be biopsied at any time point prior to study registration, bone marrow must be done at the time of study registration.

Sites of Disease: MIBG Uptake Patients must have evidence of MIBG uptake into tumor at ≥ 1 site (bone or soft tissue) within 21 days prior to study entry and subsequent to any intervening therapy. See exclusion criteria.

Autologous peripheral blood stem cells (PBSC)

* The minimum dose for peripheral blood stem cells is 1.5 x 106 viable CD34+ cells/kg. Patients who do not meet this minimum requirement for available PBSCs are not eligible.
* Only un-purged stem cells are allowed unless a center has separate FDA approval for infusion of purged stem cells.
* For patients whose body weight exceeds ideal body weight (IBW) by more than 20%, adjusted body weight may be used for the calculation of PBSC dose.47

Performance level Patients must have a Lansky (≤ 16 years) or Karnofsky (> 16 years) score of ≥ 50 Note: Subjects who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.

Prior Therapy Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to study registration.

Organ Function Requirements

Hematologic Function:

Patients must meet the following hematologic criteria for enrollment regardless of bone marrow disease involvement:

1. ANC ≥750/uL (no short-acting hematopoietic growth factors ≤ 7 days of blood draw documenting eligibility and no long-acting hematopoietic growth factors ≤ 14 days of blood draw documenting eligibility); and
2. Platelet count ≥ 50,0000/µl, transfusion independent (no platelet transfusions or platelet growth factors ≤ 7 days of blood draw documenting eligibility).

Renal Function a. Patients must have adequate renal function defined as age-adjusted serum creatinine ≤1.5 ULN for age Liver Function

1. Total bilirubin ≤ 1.5 x ULN for age; and,
2. SGPT (ALT) ≤ 135 U/L (≤ 3x ULN). Note that for ALT, the upper limit of normal for all sites is defined as 45 U/L.

Central Nervous System (CNS) Function:

1. Patients with a history of intraparenchymal or leptomeningeal based CNS disease must have no clinical or radiological evidence of active CNS disease at the time of study enrollment.
2. Patients with skull based tumors with direct intracranial extension are eligible as long as there are no neurologic signs or symptoms related to the lesion.

Cardiac Function

1. Normal ejection fraction (≥ 55%) documented by either echocardiogram or radionuclide MUGA evaluation OR normal fractional shortening (≥ 27%) documented by echocardiogram.
2. Corrected QT (QTcF) interval ≤ 480 msec. Pulmonary Function No evidence of dyspnea at rest, no exercise intolerance, or oxygen requirement. Reproductive Function

a. All females of childbearing potential (female patients 10 and older without documented ovarian failure) must have a negative serum or urine beta-HCG ≤ 7 days prior to registration.

b. Male and female subjects of reproductive age and childbearing potential must agree to use two acceptable methods of birth control (i.e., intra-uterine device, hormonal contraception, diaphragm with spermicide, condom with spermicide, or abstinence) or to abstain from heterosexual intercourse for the duration of their participation in the study, or for 3 months after last dose of protocol therapy, whichever is longer.

Exclusion Criteria:

Pregnancy, breast feeding, or unwillingness to use effective contraception during the study will not be entered on this study due to risks of fetal and teratogenic adverse events.

Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring or radiation isolation requirements of the study.

Patients with disease of any major organ system that would compromise their ability to withstand therapy.

Patients must not have received prior allogeneic stem cell transplant.

Patients who have received prior solid organ transplantation.

Patients must not have received prior total body irradiation.

Patients who are on hemodialysis.

Patients with an active or uncontrolled infection. Patients on prolonged antifungal therapy are still eligible if they are culture negative, afebrile, and meet other organ function criteria.

Known history of active human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C. Testing is not required in the absence of clinical findings or suspicion.

Patients with a history of having to permanently discontinue anti-GD2 antibody therapy, GM-CSF, or vorinostat due to toxicity are not eligible.

Patients who have received prior MIBG in combination with anti-GD2 monoclonal antibody and/or histone deacetylase inhibitor

The maximum total allowable dose of 131I-MIBG that can be given per institutional guidelines must be at least 90% of the calculated or protocol maximum 131I-MIBG dose or the patient is not eligible.

Patients with a history of deep venous thrombosis that was not associated with the presence of a central venous catheter.

Patient declines participation in NANT 2004-05, the NANT Biology Study.

Patients with evidence of active MIBG non-avid disease; patients with previously treated and stable disease that is not MIBG avid are still eligible.

Patients whose best response post previous MIBG therapy was progressive disease.

Patients with a cumulative lifetime dose of 131I-MIBG greater than 20 mCi/kg.

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 118 (Estimated)
Dates: Start 2026-07-31 (Estimated); Primary Completion 2030-07-31 (Estimated); Study Completion 2031-07-31 (Estimated)

PRIMARY OUTCOMES:
Objective Tumor Response After One Course of Therapy | 43-50 days from study day 1
  To identify the MIBG treatment regimen associated with the highest overall response rate after one course of treatment on the three arms. The response evaluation was based on central review (intent to treat analysis). Responders defined as meeting CR/MRD/PR criteria. Response was based on NANT response criteria v1.2 (https://doi.org/10.1002/pbc.26940). RECST 1.1 criteria was used for measurable tumors with PR criteria > 30% decrease in target tumor size. Curie score was used with PR criteria > 50% decrease in Curie score. Complete Response- disappearance of all target lesions, Curie score of 0 and no detectable bone marrow disease. Overall Response (OR)=CR+PR.

SECONDARY OUTCOMES:
Number of Participants With Grade 3 or Greater Non-hematologic Toxicities | All toxicities from enrollment through 30 days following end of protocol therapy, an average of 6 months
  Compare toxicity profiles for grade 3 or greater toxicities associated with each of 131I-MIBG treatment regimens; 131I-MIBG with vorinostat; 131I-MIBG with dinutuximab; or 131I-MIBG with vorinostat and dinutuximab
Objective Tumor Response After Two Courses of Therapy | 43-50 days from study day 1
  To identify the MIBG treatment regimen associated with the highest overall response rate after two courses of treatment on the three arms. The response evaluation was based on central review (intent to treat analysis). Responders defined as meeting CR/MRD/PR criteria. Response was based on NANT response criteria v1.2 (https://doi.org/10.1002/pbc.26940). RECST 1.1 criteria was used for measurable tumors with PR criteria > 30% decrease in target tumor size. Curie score was used with PR criteria > 50% decrease in Curie score. Complete Response- disappearance of all target lesions, Curie score of 0 and no detectable bone marrow disease. Overall Response (OR)=CR+PR.
Objective Bone Marrow Tumor Response After One Course of Therapy | 43-50 days from study day 1
  To identify the MIBG treatment regimen associated with the highest bone marrow response rate after one course of treatment on the three arms. The response evaluation was based on central review (intent to treat analysis). Responders defined as meeting CR/MRD/PR criteria. Response was based on NANT response criteria v1.2 (https://doi.org/10.1002/pbc.26940). RECST 1.1 criteria was used for measurable tumors with PR criteria > 30% decrease in target tumor size. Curie score was used with PR criteria > 50% decrease in Curie score. Complete Response- disappearance of all target lesions, Curie score of 0 and no detectable bone marrow disease. Overall Response (OR)=CR+PR.
Objective Bone Marrow Tumor Response After Two Courses of Therapy | 43-50 days from study day 1
  To identify the MIBG treatment regimen associated with the highest bone marrow response rate after two courses of treatment on the three arms. The response evaluation was based on central review (intent to treat analysis). Responders defined as meeting CR/MRD/PR criteria. Response was based on NANT response criteria v1.2 (https://doi.org/10.1002/pbc.26940). RECST 1.1 criteria was used for measurable tumors with PR criteria > 30% decrease in target tumor size. Curie score was used with PR criteria > 50% decrease in Curie score. Complete Response- disappearance of all target lesions, Curie score of 0 and no detectable bone marrow disease. Overall Response (OR)=CR+PR.
Objective Soft Tissue Tumor Response After One Course of Therapy | 43-50 days from study day 1
  To identify the MIBG treatment regimen associated with the highest soft tissue response rate after one course of treatment on the three arms. The response evaluation was based on central review (intent to treat analysis). Responders defined as meeting CR/MRD/PR criteria. Response was based on NANT response criteria v1.2 (https://doi.org/10.1002/pbc.26940). RECST 1.1 criteria was used for measurable tumors with PR criteria > 30% decrease in target tumor size. Curie score was used with PR criteria > 50% decrease in Curie score. Complete Response- disappearance of all target lesions, Curie score of 0 and no detectable bone marrow disease. Overall Response (OR)=CR+PR.
Objective Soft Tissue Tumor Response After Two Courses of Therapy | 43-50 days from study day 1
  To identify the MIBG treatment regimen associated with the highest soft tissue response rate after two courses of treatment on the three arms. The response evaluation was based on central review (intent to treat analysis). Responders defined as meeting CR/MRD/PR criteria. Response was based on NANT response criteria v1.2 (https://doi.org/10.1002/pbc.26940). RECST 1.1 criteria was used for measurable tumors with PR criteria > 30% decrease in target tumor size. Curie score was used with PR criteria > 50% decrease in Curie score. Complete Response- disappearance of all target lesions, Curie score of 0 and no detectable bone marrow disease. Overall Response (OR)=CR+PR.
Objective Bone Tumor Response After One Course of Therapy | 43-50 days from study day 1
  To identify the MIBG treatment regimen associated with the highest bone response rate after one course of treatment on the three arms. The response evaluation was based on central review (intent to treat analysis). Responders defined as meeting CR/MRD/PR criteria. Response was based on NANT response criteria v1.2 (https://doi.org/10.1002/pbc.26940). RECST 1.1 criteria was used for measurable tumors with PR criteria > 30% decrease in target tumor size. Curie score was used with PR criteria > 50% decrease in Curie score. Complete Response- disappearance of all target lesions, Curie score of 0 and no detectable bone marrow disease. Overall Response (OR)=CR+PR.
Objective Bone Tumor Response After Two Courses of Therapy | 43-50 days from study day 1
  To identify the MIBG treatment regimen associated with the highest bone response rate after two courses of treatment on the three arms. The response evaluation was based on central review (intent to treat analysis). Responders defined as meeting CR/MRD/PR criteria. Response was based on NANT response criteria v1.2 (https://doi.org/10.1002/pbc.26940). RECST 1.1 criteria was used for measurable tumors with PR criteria > 30% decrease in target tumor size. Curie score was used with PR criteria > 50% decrease in Curie score. Complete Response- disappearance of all target lesions, Curie score of 0 and no detectable bone marrow disease. Overall Response (OR)=CR+PR.
Objective MIBG Tumor Response After One Course of Therapy | 43-50 days from study day 1
  To identify the MIBG treatment regimen associated with the highest MIBG response rate after one course of treatment on the three arms. The response evaluation was based on central review (intent to treat analysis). Responders defined as meeting CR/MRD/PR criteria. Response was based on NANT response criteria v1.2 (https://doi.org/10.1002/pbc.26940). RECST 1.1 criteria was used for measurable tumors with PR criteria > 30% decrease in target tumor size. Curie score was used with PR criteria > 50% decrease in Curie score. Complete Response- disappearance of all target lesions, Curie score of 0 and no detectable bone marrow disease. Overall Response (OR)=CR+PR.
Objective MIBG Tumor Response After Two Courses of Therapy | 43-50 days from study day 1
  To identify the MIBG treatment regimen associated with the highest MIBG response rate after two courses of treatment on the three arms. The response evaluation was based on central review (intent to treat analysis). Responders defined as meeting CR/MRD/PR criteria. Response was based on NANT response criteria v1.2 (https://doi.org/10.1002/pbc.26940). RECST 1.1 criteria was used for measurable tumors with PR criteria > 30% decrease in target tumor size. Curie score was used with PR criteria > 50% decrease in Curie score. Complete Response- disappearance of all target lesions, Curie score of 0 and no detectable bone marrow disease. Overall Response (OR)=CR+PR.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Children Hospital of Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Childrens Hospital Boston, Dana-Farber Cancer Institute., Boston, Massachusetts
  - C.S Mott Children's Hospital, Ann Arbor, Michigan
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided